CLINICAL TRIAL: NCT04292587
Title: Prevalence of Hirsutism in Turkey: Data of The Dermatoendocrinology Study Group
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Filiz Cebeci Kahraman, Associate Professor, Istanbul Medeniyet University
Other Study IDs: 08122018
Record Dates: First submitted 2020-02-26; First posted 2020-03-03 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Hirsutism
Keywords: Ferriman-Gallwey score, hirsutism, prevalence
MeSH Terms: conditions — Hirsutism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women with hirsutism: Women between the ages of 18-45 with hirsutism
- Women without hirsutism: Women between the ages of 18-45 without hirsutism

SUMMARY:
Hirsutism is defined as the excessive presence of terminal hairs in the androgen-sensitive areas of the female body, and it is one of the frequent reasons for presenting to dermatology outpatient clinics. Hirsutism influences 5% to 10% of women around the world and leads to psychological problems depending on ethnic and socio-cultural factors. It also causes material burden including medicines, cosmetic products and epilation procedures.

The differences in the real prevalence of hirsutism in the Turkish population and the hirsutism prevalence and severity between the geographical regions of Turkey are not known. In this study, we aimed to determine the prevalence of hirsutism in women at the reproductive age within Turkey. The geographical regions of Turkey comprise seven regions and and all regions were included in this study. By considering the regions where ethnic differences were high including the east-west-south and north of our country, we aimed to find an answer to the question of whether there were differences in terms of the prevalence and severity of hirsutism among these regions. A comprehensive study aiming to determine the prevalence of hirsutism in Turkey has not been conducted.

DETAILED DESCRIPTION:
Twenty-two provinces of Turkey's seven regions and 26 hospitals from these provinces will be included in the study. The number of samples was specified by the public health specialist on the 2018 census figures. The Turkish population consists of 80,810,525 people according to the data announced by the Turkish Statistical Institute in 2018. In order to determine the prevalence in Turkey, the sample size was calculated with a confidence interval of 99% and error margin of 1%, and the total number of individuals to be screened was designated as 5861. The number of patients to be screened via the clustering method weighted by regions was specified as 1800 for the Marmara Region, 750 for the Aegean Region, 744 for the Mediterranean Region, 568 for the Black Sea Region, 932 for the Central Anatolia Region, 434 for the Eastern Anatolia Region and 633 for the Southeastern Anatolia Region. The provinces that were thought to represent each region were selected via the cluster sampling method.

During the study period, female patients aged between 18 and 45, who present to dermatology outpatient clinics, will be examined clinically until the number of patients designated for each study center is reached, and the hirsutism level of the patients diagnosed with hirsutism will be determined by using the modified Ferriman-Gallwey (mFG) scoring system. In this system, hair growth in nine regions (upper lip, chin, chest, upper back, lower back, upper abdomen, lower abdomen, upper arms and thighs) is graded between 0 and 4. And nine regions are scored between 0 (no terminal hairs) and 4 (excessive presence of terminal hairs). The score above 8 is considered hirsutism. The hirsutism family history, body mass index, menstrual cycle pattern, concomitant disease status (diabetes, hyperlipidemia, hypertension, thyroid disease), history of medication causing body hair growth, the acne presence and severity, presence and severity of androgenic alopecia, presence of seborrhea, presence and localization of acanthosis nigricans, presence of acrochordon, presence of hidradenitis suppurativa, presence of galactorrhea, presence of virilization symptoms and presence of cushingoid symptoms of all the examined patients will be investigated and recorded.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged between 18 and 45, who presented to the dermatology outpatient clinics for any reason
* Not being in pregnancy and lactation period
* Not applying permanent epilation
* Not using temporary hair reduction methods in the last 4 weeks
* Not using oral contraceptive, corticosteroid, cyclosporin or spironolactone in the last 3 months

Exclusion Criteria:

* Female patients below the age of 18, above 45 and men in any age group
* Pregnant women and women in lactation period
* Patients who had permanent epilation
* Patients who had temporary hair reduction methods in the last 4 weeks
* Patients taking oral contraceptive, corticosteroid, cyclosporin or spironolactone in the last 3 months

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: During the study period, female patients aged between 18 and 45, who present to dermatology outpatient clinics, will be examined consecutive until the number of patients designated for each study center is reached.
Sampling Method: Probability Sample
Enrollment: 5861 (Estimated)
Dates: Start 2020-02-03 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Modified Ferriman-Gallwey Scoring System for Severity of Hirsutism | 1 day (At the time of the examination)
  In this system, hair growth in nine regions (upper lip, chin, chest, upper back, lower back, upper abdomen, lower abdomen, upper arms and thighs) is graded between 0 and 4. And nine regions are scored between 0 (no terminal hairs) and 4 (excessive presence of terminal hairs). The score above 8 is considered hirsutism.

SECONDARY OUTCOMES:
Number of Participants With Concomitant disease status and the risk factors | 1 day (At the time of the examination)
  Concomitant disease status (diabetes, hyperlipidemia, hypertension, thyroid disease), hirsutism family history, history of medication causing body hair growth, presence of seborrhea, presence and localization of acanthosis nigricans, presence of acrochordon, presence of hidradenitis suppurativa, presence of galactorrhea, presence of virilization symptoms and presence of cushingoid symptoms of all the examined patients will be determined and recorded.
Body mass indices of the participants | 1 day (At the time of the examination)
  BMI in kg/m^2
The presence and severity of acne in the participants | 1 day (At the time of the examination)
  If acne is present, it will be classified as mild, moderate and severe.
The presence and severity of androgenic alopecia in the participants | 1 day (At the time of the examination)
  If androgenic alopecia is present, it will be classified as Ludwig 1, Ludwig 2, Ludwig 3.
Menstrual cycle pattern of the participants | 1 day (At the time of the examination)
  The menstrual cycle pattern of the participants will be classified as regular, oligomenorrhea, amenorrhea, polimenorrhea

CONTACTS AND LOCATIONS:
Overall Officials: Filiz Cebeci Kahraman, Assoc. Prof., Principal Investigator — University of Health Sciences, Goztepe Training and Research Hospital
Locations (26):
- Turkey (Türkiye) (26):
  - Adana City Training and Research Hospital, Adana
  - School of Medicine, Aksaray University, Aksaray
  - School of Medicine, Ankara Yıldırım Beyazıt University, Ankara
  - School of Medicine, Aydın Adnan Menderes University, Aydin
  - Bitlis Tatvan State Hospital, Bitlis
  - School of Medicine, Uludag University, Bursa
  - University of Health Sciences, Gazi Yasargil Training and Research Hospital, Diyarbakır
  - School of Medicine, Trakya University, Edirne
  - School of Medicine, Eskisehir Osmangazi University, Eskişehir
  - School of Medicine, Gaziantep University, Gaziantep
  - School of Medicine, Süleyman Demirel University, Isparta
  - University of Health Sciences, Bakırköy Sadi Konuk Training and Research Hospital, Istanbul
  - University of Health Sciences, Sultan 2. Abdulhamid Han Training and Research Hospital, Istanbul
  - Istanbul Medeniyet University, Goztepe Research and Training Hospital, Istanbul
  - University of Health Sciences, Umraniye Training and Research Hospital, Istanbul
  - Marmara University Pendik Training and Research Hospital, Istanbul
  - School of Medicine,Izmir Katip Celebi University, Izmir
  - School of Medicine,Kahramanmaras Sutcu Imam University, Kahramanmaraş
  - School of Medicine, Kocaeli University, Kocaeli
  - Meram School of Medicine, Necmettin Erbakan University, Konya
  - School of Medicine, Celal Bayar University, Manisa
  - Sanlıurfa Training and Research Hospital, Sanliurfa
  - School of Medicine, Namık Kemal University, Tekirdağ
  - School of Medicine,Tokat Gaziosmanpasa University, Tokat Province
  - School of Medicine,Karadeniz Technical University, Trabzon
  - University of Health Sciences, Van Training and Research Hospital, Van

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li R, Qiao J, Yang D, Li S, Lu S, Wu X, Wei Z. Epidemiology of hirsutism among women of reproductive age in the community: a simplified scoring system. Eur J Obstet Gynecol Reprod Biol. 2012 Aug;163(2):165-9. doi: 10.1016/j.ejogrb.2012.03.023. Epub 2012 Jun 28. PMID 22748844
- [Background] Lumezi BG, Berisha VL, Pupovci HL, Goci A, Hajrushi AB. Grading of hirsutism based on the Ferriman-Gallwey scoring system in Kosovar women. Postepy Dermatol Alergol. 2018 Dec;35(6):631-635. doi: 10.5114/ada.2018.77615. Epub 2018 Nov 13. PMID 30618534
- [Background] Fatemi Naeini F, Najafian J, Jazebi N. Hirsutism and body mass index in a representative sample of Iranian people. ARYA Atheroscler. 2012 Spring;8(1):43-54. PMID 23056100
- [Background] Carmina E. Prevalence of idiopathic hirsutism. Eur J Endocrinol. 1998 Oct;139(4):421-3. doi: 10.1530/eje.0.1390421. PMID 9820619